CLINICAL TRIAL: NCT01954589
Title: Double-blind, Placebo- and Active-controlled, Randomized, Single-ascending Dose Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of ACT-462206 in Healthy Male Subjects
Brief Title: Single-ascending Dose Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of ACT-462206
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AC-074-101
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Safety; Tolerability; Pharmacodynamics; Pharmacokinetics
Keywords: ACT-462206; Selective dual orexin receptor antagonist
MeSH Terms: interventions — ACT-462206; almorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- ACT-462206 5 mg/Placebo (Experimental): 6 subjects received a single, 5 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 5 mg; Drug: Placebo
- ACT-462206 25 mg/Placebo (Experimental): 6 subjects received a single, 25 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 25 mg; Drug: Placebo
- ACT-462206 100mg/Placebo (Experimental): 6 subjects received a single, 100 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 100mg; Drug: Placebo
- ACT-462206 200mg/Almorexant 400mg/Placebo (Experimental): Subjects were assigned to one of two possible treatment sequences: A/B or B/A with a washout period of 14 days between treatment periods.
  Treatment A: Single oral dose of ACT-462206 200 mg or placebo. Treatment B: Single oral dose of almorexant 400 mg or placebo. In each sequence 6 subjects received ACT-462206 or almorexant & 2 subjects received placebo
  Interventions: Drug: ACT-462206 200mg; Drug: Almorexant 400mg; Drug: Placebo
- Experimental: ACT-462206 400mg/Placebo (Experimental): 6 subjects received a single, 400 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 400mg; Drug: Placebo
- ACT-462206 1000 mg (Experimental): 6 subjects received a single, 1000 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 1000 mg; Drug: Placebo
- ACT-462206 1500mg/Placebo (Experimental): 6 subjects received a single, 1500 mg, oral dose of ACT-462206 and 2 subjects received a single, oral dose of placebo
  Interventions: Drug: ACT-462206 1500mg; Drug: Placebo

INTERVENTIONS:
Drug: ACT-462206 5 mg
  Arms: ACT-462206 5 mg/Placebo
Drug: ACT-462206 25 mg
  Arms: ACT-462206 25 mg/Placebo
Drug: ACT-462206 100mg
  Arms: ACT-462206 100mg/Placebo
Drug: ACT-462206 200mg
  Arms: ACT-462206 200mg/Almorexant 400mg/Placebo
Drug: ACT-462206 400mg
  Arms: Experimental: ACT-462206 400mg/Placebo
Drug: ACT-462206 1000 mg
  Arms: ACT-462206 1000 mg
Drug: ACT-462206 1500mg
  Arms: ACT-462206 1500mg/Placebo
Drug: Almorexant 400mg
  Arms: ACT-462206 200mg/Almorexant 400mg/Placebo
Drug: Placebo

SUMMARY:
A study of ACT-462206 to evaluate the tolerability, safety, pharmacokinetics, and pharmacodynamic of ascending single doses of ACT-462206, a novel dual orexin receptor antagonist in healthy male subjects.

DETAILED DESCRIPTION:
Each dose level will be investigated in a new group of eight healthy male subjects (six on active drug and two on placebo). Each subject will participate in one treatment period, with the exception of subjects in the crossover part (i.e., almorexant reference group at the fourth dose level), who will participate in two treatment periods. At this dose level subjects on active drug (six) will receive in one treatment period ACT-462206 and in the other 400 mg of almorexant; subjects on placebo (two) will receive the corresponding placebos (double-dummy).

ELIGIBILITY:
Inclusion Criteria

* Healthy male subjects aged between 18 and 45 years (inclusive) at screening
* Hematology, clinical chemistry, and urinalysis results not deviating from the normal range to a clinically relevant extent at screening
* No clinically significant findings on physical examination at screening
* Body mass index between 18.0 and 28.0 kg/m^2 (inclusive) at screening
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and heart rate 45-90 beats per minute (inclusive) measured at screening on the dominant arm (dominant arm is the writing arm) after 5 min in supine position
* 12-lead electrocardiogram without clinically relevant abnormalities in the supine position at screening
* Negative results from urine drug screen at screening
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Treatment with any prescribed medications (including vaccines) or over-the-counter medications (including herbal medicines such as St John's Wort) within 2 weeks prior to (first) study drug administration
* Treatment with another investigational drug within 3 months prior to screening or having participated in more than four investigational drug studies within 1 year prior to screening
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening
* History or clinical evidence of any disease, and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening of caffeine)
* Smoking within 3 months prior to screening and inability to refrain from smoking during the course of the study
* Loss of 250 mL or more of blood, or an equivalent amount of plasma, within 3 months prior to screening
* Positive results from the hepatitis serology, except for vaccinated subjects or subjects with past but resolved hepatitis, at screening
* Positive results from the human immunodeficiency virus serology at screening
* Known hypersensitivity to any excipients of the drug formulations
* Modified Swiss Narcolepsy Scale total score < 0 or history of narcolepsy or cataplexy
* Any circumstances or conditions, which, in the opinion of the investigator, might affect full participation in the study or compliance with the protocol
* Legal incapacity or limited legal capacity at screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in supine systolic blood pressure from baseline up to the end of study | 96 hours
  Blood pressure was measured on the dominant arm using an automatic oscillometric device. Measurements were taken with the subject in the supine position after a resting period of at least 5 min. The dominant (writing) arm was used for all measurements. Measurements were taken at 1, 3, 5, 8, 24, 48, 72 and 96 hours post-dose.
Change in supine diastolic blood pressure from baseline up to the end of study | 96 hours
  Blood pressure was measured on the dominant arm using an automatic oscillometric device. Measurements were taken with the subject in the supine position after a resting period of at least 5 min. The dominant (writing) arm was used for all measurements. Measurements were taken at 1, 3, 5, 8, 24, 48, 72 and 96 hours post-dose.
Change in heart rate from baseline up to the end of study | 96 hours
  Heart rate was measured on the dominant arm using an automatic oscillometric device. The dominant (writing) arm was used for all measurements. Measurements were taken at 1, 3, 5, 8, and 96 hours post-dose.
Change in body weight from baseline up to the end of study | 96 hours
  Body weight will be measured using the same weighing scale for all subjects and throughout the study. The weighing scale should have a precision of at least 0.5 kg.
Change in PR Interval from baseline up to the end of study | 96 hours
  A standard 12-lead electrocardiogram (ECG) was recorded in supine position after a 5-min rest period. The PR interval is the time interval from the beginning of the P wave to the beginning of the QRS complex. Measurements were taken at 1, 3, 5, 8, and 96 hours post-dose.
Change in QRS Interval from baseline up to the end of study | 96 hours
  A standard 12-lead ECG was recorded in supine position after a 5-min rest period. The QRS interval is the time interval from the beginning of the Q wave to the end of the S wave. Measurements were taken at 1, 3, 5, 8, and 96 hours post-dose.
Change in QTcB Interval from baseline up to the end of study | 96 hours
  A standard 12-lead ECG was recorded in supine position after a 5-min rest period. The QTcB interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate). Measurements were taken at 1, 3, 5, 8, and 96 hours post-dose.
Change in QTcF Interval from baseline up to the end of study | 96 hours
  A standard 12-lead ECG was recorded in supine position after a 5-min rest period. The QTcF interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Fridericia's formula (QTcF = QT/RR^0.33 where RR is 60/heart rate). Measurements were taken at 1, 3, 5, 8, and 96 hours post-dose.
Change in saccadic peak velocity from baseline up to the end of study | 10 hours
  Recording of eye movements was performed in a quiet room with ambient illumination, with only 1 subject present. A microcomputer system was used for recording & analysis. Disposable electrodes were applied on the forehead & beside the lateral canthi of both eyes for registration of the electro-oculographic signals. Head movements were restricted using a fixed head support. The target consisted of a moving dot displayed on a computer screen, fixed in front of the head support. Saccadic eye movements were recorded for stimulus amplitudes of approximately 15 degrees to either side. Fifteen saccades were recorded with inter-stimulus intervals varying randomly between 3 and 6 s. Average values of saccadic peak velocity of all correct saccades were used as variables.Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.
Change in performance on adaptive tracking from baseline up to the end of study | 10 hours
  The adaptive tracking test was performed using customized equipment and software, following a standard protocol. Adaptive tracking is a pursuit-tracking task. The subject was asked to keep a dot inside a randomly moving circle by operating a joystick. If successful, the speed of the moving circle was increased. Conversely, the velocity was reduced if the subject could not maintain the dot inside the circle. The average performance (%) and the standard deviation of scores during a 3.5-min assessment period were used for analysis. The assessment period included a run-in time of 0.5 min, during which data were not recorded.Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.
Change in body sway from baseline up to the end of study | 10 hours
  Body sway was assessed using a body sway meter. All body movements during a 2-min period of time were integrated and expressed as mm sway on a digital display. Measurements of body sway were made in the sagittal (forward/backward) planes by positioning of the subject relative to the apparatus, with a string attached to the waist. The contribution of vision to postural control was eliminated by asking subjects to close their eyes. Subjects were instructed to wear the same pair of comfortable, low-heeled shoes in each session. Before starting a measurement, subjects were asked to stand still and comfortable, with their feet approximately 10 cm apart and their hands in a relaxed position alongside the body. Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.
Change in visual analogue scale (VAS) score to assess alertness from baseline up to the end of study | 10 hours
  Dutch versions of the VAS according to Bond and Lader (British Journal of Medical Psychology 1974;47:211-18) were used to assess subjective alertness. At each time point of assessment, the subject indicated (with a mouse click on the computer screen) how he felt, on sixteen dimension horizontal VAS. Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.
Change in VAS score to assess mood from baseline up to the end of study | 10 hours
  Dutch versions of the VAS according to Bond and Lader (British Journal of Medical Psychology 1974;47:211-18) were used to assess subjective mood. At each time point of assessment, the subject indicated (with a mouse click on the computer screen) how he felt, on sixteen dimension horizontal VAS. Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.
Change in VAS score to assess calmness from baseline up to the end of study | 10 hours
  Dutch versions of the VAS according to Bond and Lader (British Journal of Medical Psychology 1974;47:211-18) were used to assess subjective calmness. At each time point of assessment, the subject indicated (with a mouse click on the computer screen) how he felt, on sixteen dimension horizontal VAS. Measurements were taken at 20 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, and 10 hours post-dose.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-462206 | 96 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours after dosing. Cmax calculated on the basis of the blood sampling time points.
Time to reach maximum plasma concentration (tmax) of ACT-462206 | 96 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours after dosing. tmax calculated on the basis of the blood sampling time points.
Area under the plasma concentration-time curve (AUC) from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) of ACT-462206 | 96 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours after dosing. AUC0-t was calculated on the basis of the blood sampling time points, according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.
AUC from time zero to infinity (AUC0-∞) of ACT-462206 | 96 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours after dosing. AUC0-∞ was calculated by combining AUC0-t and AUCextra. AUCextra is an extrapolated value obtained by Ct/λz, where Ct is the last plasma concentration measured above the limit of quantification and λz represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations in the terminal elimination phase.
AUC from time zero to 8 hours after administration (AUC0-8) of ACT-462206 | 8 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, and 8 hours, after dosing. AUC0-8 was calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.
AUC from time zero to 24 hours after administration (AUC0-24) of ACT-462206 | 24 hours
  Blood samples for pharmacokinetic analysis taken immediately prior to dosing with ACT-462206, and at 10 minutes, 20 minutes, 30 minutes, 45 minutes, 60 minutes, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, and 24 hours after dosing. AUC0-24 was calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Baecker, MD, Study Director — Actelion
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands